CLINICAL TRIAL: NCT06080126
Title: Developing and Implementing Meaningful Activities Facilitators in Short-stay Geriatric Unit to Prevent Geriatric Complication - A Feasibility Study
Brief Title: Developing and Implementing Meaningful Activities Facilitators in Geriatric Short Stay
Acronym: MAYFAIR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL22_0726; 2023-A00490-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2023-09-21; First posted 2023-10-12 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Geriatric Care
Keywords: Meaningful activities facilitators; geriatric service

STUDY DESIGN:
Intervention Model Description: The study will be conducted in a 2-phase approach corresponding to the 2 successive phases of the MRC guidance:
  * Phase 1: The adaptation of the intervention to our context will be based on a literature review and a qualitative study.
  * Phase 2: The feasibility and acceptability of the intervention will be assessed during a quasi-experimental before and after study conducted in two short-stay geriatric units.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other)
  Interventions: Other: Control: per usual practice
- Intervention (Other)
  Interventions: Other: Intervention MAF

INTERVENTIONS:
Other: Control: per usual practice — 160 patients were included as per usual practice.
  Arms: Control
Other: Intervention MAF — 160 patients were included with MAF intervention.
  Arms: Intervention

SUMMARY:
Older people are particularly vulnerable to adverse effects of hospitalization, which can compromise their functional autonomy. The onset of confusion, loss of mobility or malnutrition is largely related to the context of hospitalization itself, which creates stressful situations for patients in addition to the acute pathology: change in the usual living environment, lack of human and reassuring interactions, lack of mobility related to the pathology or caused by the use of barriers or restraints. These geriatric complications can be prevented. Programs involving the intervention of volunteers or dedicated professionals with hospitalized patients have been developed. These "Meaningful Activities Facilitators" (MAF) have the task of preventing or limiting the deleterious effects of hospitalization on the older people, in particular by stimulating eating and walking, and by practicing social activities in line with the patient's lifestyle habits. This system has been set up in geriatric short-stay wards in the United Kingdom, where MAFs, who received specific training, are integrated into the care team and work with patients at risk. The integration of these MAFs has shown a reduction in the incidence and duration of delirium episodes, the use of psychotropic drugs, and the use of restraint. A study currently underway in Australia aims to reduce hospital-acquired complications through a program of mobilization, nutrition, and engagement of patients in constructive activities (the "Eat, Walk, Engage" program) implemented by a trained MAFs. The investigators hypothesis is that the implementation of MAFs in geriatric short-stay wards will reduce the incidence of geriatric complications associated with hospitalization.

Objectives: The investigators objective is to study the feasibility and acceptability of integrating MAFs into the care teams of two geriatric short-stay services in France. The investigators will evaluate the adaptations to be proposed to the MAF model to make it relevant in our context from the point of view of patients, their relatives and professionals, and will study the effect of this intervention on the occurrence of complications and the functioning of the teams, its implementation and its costs.

Perspectives: The results of this study will allow us to define if the MAFs intervention is feasible and acceptable in the French context, and if so, to propose an intervention model adapted to our context.

DETAILED DESCRIPTION:
Methods: The project will be carried out in 2 phases guided by the Medical Research Council's (MRC) recommendations for the development and evaluation of complex health interventions. Phase 1: Adaptation of the MAFs intervention to our context, combining literature review, non-participant observation, semi-structured interviews, and coconstruction workshops. Phase 2: Feasiblity testing : A quasi-experimental feasibility "before and after" study will be conducted in two geriatric short-stay services on 380 patients: "before" period over 4 months (inclusion of 160 hospitalized patients constituting the control group), recruitment and training of 2 MAFs, implementation of the intervention, "after" period over 4 months (inclusion of 160 hospitalized patients constituting the intervention group). The patients will be included at admission and followed up during the hospital stay. The data collected concern the occurrence of complications during the stay, the quality of life at work of the professionals, and in the "after" period, the acceptability and fidelity of the MAFs intervention, according to the point of view of the MAFs, the professionals and the patients/relatives. These criteria will be collected through monitoring of the MAFs activity (logbook, medical records) and semi-structured interviews. The impact of the integration of the MAFs on the functioning, team cohesion and collaboration will be studied.

The results will allow us to propose phase 3 of the MRC recommendations, a multicenter randomized controlled evaluation in clusters, informed by the results for the content of the intervention, the implementation strategies, the choice of the primary endpoint, the inclusion criteria of the population, the calculation of the sample size and the study procedures (inclusion, data collection).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 and over
* admitted to a geriatric short-stay hospital for > 72 hours
* Considered "at risk of complications related to hospitalisation": at least two of the following criteria:

  * Clinical Frailty Scale (Rockwood Clinical Frailty Score
  * At least one ADL-IADL dependency,
  * Presence of known cognitive impairment,
  * Patient confused on admission,
  * History of confusional syndrome on previous hospitalisation or use of medication,
  * Anxiety-depression (history or current pathology),
  * Repeated falls (>2 in a year) or fear of falling,
  * Risk of sarcopenia (Score >4 on the SARC-F questionnaire
  * Presenting undernutrition or a risk of undernutrition (according to medical assessment, e.g. low BMI, anorexia, recent weight loss).
* Patient having been informed of the study and having signed an informed consent (for patients under guardianship, the consent of the guardian will be requested). For patients under guardianship, the patient will sign the consent in the presence of the guardian.
* Patient who understands and speaks French
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Patient in palliative care for a terminal disease
* Re-hospitalised patients already included during a previous stay
* Patients under court protection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of implementing meaningful activities facilitators (MAF) in a French short stay geriatric unit, from the perspective of professionals, MAF and patients/relatives. | From the implementation of a meaningful activities facilitators for a period of 4 months.
  Criteria to conclude on feasibility will be the fulfilment of the following criteria during the intervention period (MAF implementation):
  * employment of two MAFs (one per participating unit, 0.5FTE),
  * SATIN and EEPMT Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Geriatric Short Stay Department - Unit 3C of the Charpennes Hospital, Lyon
  - University Department of Geriatric Medicine, Centre Hospitalier Lyon Sud, Lyon

IPD SHARING:
Plan to Share IPD: No